CLINICAL TRIAL: NCT02716935
Title: Effect of Supplementation With LNS Fortified With a Mixture of FOS and Inulin on Gut Microbiota Diversity and Functionality and Its Repercussion on Growth and Morbidity During Infancy in Rural Burkina Faso
Brief Title: Prebiotics and Microbiota Composition and Functionality in Rural Burkinabe Infants
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Ghent (Other)
Collaborators: Institut de Recherche en Sciences de la Sante, Burkina Faso (Other Government); Nutriset (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: University Ghent
Record Dates: First submitted 2016-02-01; First posted 2016-03-23 (Estimated); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Growth Retardation; Infant Morbidity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (3):
- Fortified lipid based nutrient supplement (Experimental): lipid based nutrient supplement (Nutributter) fortified with fructo-oligosaccharides and inulin
  Interventions: Dietary Supplement: Fortified lipid based nutrient supplement
- lipid based nutrient supplement (Active Comparator): lipid based nutrient supplement (Nutributter)
  Interventions: Dietary Supplement: lipid based nutrient supplement
- non intervention group (No Intervention): This group will not be supplemented

INTERVENTIONS:
Dietary Supplement: Fortified lipid based nutrient supplement — 6 months intervention: participant will take a daily dose of 20g supplement. The product contains 3 g of a mixture (1:1) of inulin and fructan-oligosaccharide
  Arms: Fortified lipid based nutrient supplement
Dietary Supplement: lipid based nutrient supplement — Dietary Supplement: lipid based nutrient supplement (Nutributter) 6 months intervention: participant will take a daily dose of 20g supplement.
  Arms: lipid based nutrient supplement

SUMMARY:
The purpose of this study is to assess the effect of a mixture of prebiotics included in a food supplement on microbiota diversity and functionality, and to explore its subsequent effects on linear growth velocity and morbidity.

DETAILED DESCRIPTION:
The central role of gut microbiota in immunity and nutritional homeostasis is now acknowledged, albeit not fully understood. Gut microbiota composition imbalances have been found in malnourished children, which were not restored by nutritional interventions as currently conducted. Therefore, the necessity to design more complete nutritional interventions that include gut health has been advised by expert committees.

Prebiotics are compound that selectively enhance the growth of beneficial gut bacteria. They have been recommended and used in infant formula and weaning cereals resulting in gut microbiota resembling that of breastfed infants in formula fed infants in developed countries. A healthy gut microbiota was shown to be associated with enhanced growth patterns and decreased morbidity in children in developed countries. Evidence of such outcome is lacking in developing countries, yet such results would be particularly valuable for children from these settings, living in rather poor sanitary conditions in an environment characterized with high infectious disease load, conditions that mostly explain the high prevalence of chronic malnutrition. This study aims to assess the effect of a 6 months' supplementation with a lipid based nutrient supplement fortified with fructo-oligosaccharides and inulin on microbiota diversity and functionality in rural Burkinabe infants, and to explore its subsequent effects on linear growth velocity and morbidity.

ELIGIBILITY:
Inclusion Criteria:

* 6-6.5 month old infants
* Weight for height and height for age z-score above -2
* Permanent resident of the area and not intending to move for the next 6 months for more than a week
* No chronic antibiotic treatment
* Exempt of any current serious illness
* Still breastfed.

Exclusion Criteria:

* Moderate or severe malnutrition (weight for height or height for age z-score below -2)
* non-permanent residence in the study area,
* the presence of any congenital anomalies in the child or mental/physical disease of the mother that can interfere with child feeding
* a chronic antibiotic treatment i.e. more than 6 weeks treatment at the time of enrolment
* a history of allergy to a constituent of the supplement
* a serious current illness

Ages: 24 Weeks to 26 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 153 (Actual)
Dates: Start 2016-03; Primary Completion 2018-04-24 (Actual); Study Completion 2019-11 (Actual)

PRIMARY OUTCOMES:
Fecal microbiota range-weighted richness | 6 months
  Composition of fecal microbiota will be determined by Illumina sequencing from which range-weighted richness will be calculated
Mean concentration of short-chain fatty acids in stool | 6 months
  Concentration of short-chain fatty acids (acetate, butyrate and propionate) will be measured by Gas Chromatography

SECONDARY OUTCOMES:
Frequency of digestive intolerance symptoms (flatulence, abdominal pain, regurgitation, vomiting, or diarrhea) | once every week during the first month of supplementation
  Digestive intolerance symptoms will be recalled.
Stool consistency | Once every week during the first month of supplementation
  Stool consistency will be recalled
Stool frequency per day | 6 months
  Stool frequency per day will be recalled.
Mean stool pH | once every week during the first month of supplementation
  Stool pH will be measured once a week with pH sticks by a study nurse
Calprotectin concentration in stool | at inclusion, 3 months and 6months after inclusion
  Concentration of calprotectin will be measured by ELISA
Infant linear growth velocity | once a month during 6 months
  Linear growth velocity will be determined using the difference between 2 length measures over the follow up time in months and expressed in millimeters/ month
Infant ponderal growth velocity | once a month during 6 months
  Ponderal growth velocity will be determined using the difference between 2 weight measures over the follow up time in month and expressed in grams/ month. Infant's weight will be measured at inclusion and once a month during 6 months
Cumulative morbidity | Starting from inclusion, weekly during a follow-up of 6 months
  Cumulative morbidity of (malaria, gastro-intestinal tract infection, acute respiratory tract infection, acute otitis) will be assessed one a week by a study nurse
Infant's intestinal permeability | at inclusion, 3 months and 6 months after inclusion
  Intestinal permeability will be assessed using a mannitol-lactulose test
Residual fecal microbiota range-weighted richness | 3 months and 6 months
  Composition of fecal microbiota will be determined by Illumina sequencing, from which range-weighted richness will be calculated
Residual concentration of short-chain fatty acids in stool | 3 months and 6 months
  Concentration of short chain fatty acids (acetate, butyrate and propionate) will be measured by Gas Chromatography

CONTACTS AND LOCATIONS:
Locations (1):
- IRSS/DRO, Bobo-Dioulasso, Houet, Burkina Faso

IPD SHARING:
Plan to Share IPD: Yes
Upon publication of the main findings, data will be shared on a public repository and made publicly available on request as per recently published guidance and regulations (BMJ 2016;352:i255)